CLINICAL TRIAL: NCT07224893
Title: Once-Daily Versus Twice-Daily Insulin Glargine in the Management of Patients With Pregestational Diabetes Requiring Insulin
Brief Title: Once-Daily vs Twice-Daily Insulin Glargine in Pregestational Diabetes Management
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Marwan Ma'ayeh, Assistant Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-09-FB-0214
Record Dates: First submitted 2025-10-31; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Pregestational Diabetes; Pregnancy
Keywords: continuous glucose monitoring

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Once-Daily Insulin Glargine (Active Comparator): Participants randomized to this arm will take insulin glargine once daily
  Interventions: Drug: Use of insulin glargine once daily
- Twice-Daily Insulin Glargine (Experimental): Participants randomized to this arm will take insulin glargine twice daily
  Interventions: Drug: Use of insulin glargine twice daily

INTERVENTIONS:
Drug: Use of insulin glargine once daily — Insulin glargine will be used once daily
  Arms: Once-Daily Insulin Glargine
Drug: Use of insulin glargine twice daily — Insulin glargine will be used twice daily
  Arms: Twice-Daily Insulin Glargine

SUMMARY:
The purpose of this study is to determine if taking insulin glargine twice a day instead of once a day will better manage pregestational diabetes in pregnant patients. Participants in this study will be randomly assigned to one of two groups: a group that takes insulin glargine once a day, and a group that takes it twice. Continuous glucose monitoring will be used to track blood sugar levels. The main question the study aims to answer is: Will using insulin glargine twice a day instead of once lead to a better glucose time in range?

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age;
* The patient is fluent in English, physically and mentally able to understand the informed consent, and is willing to participate in this study;
* Type II diabetes mellitus requiring insulin;
* The patient is between 24 weeks 0 days and 28 weeks 0 days of gestation at the time of enrollment. Gestational age will be determined by last menstrual period, confirmed with a first trimester ultrasound, per the recommended guidelines by the American College of Obstetricians and Gynecologists.
* Currently using or willing to use a clinically indicated continuous glucose monitor for glycemic management

Exclusion Criteria:

* Known allergy or reaction to insulin glargine, or concurrent medical condition where the use of insulin glargine is contraindicated;
* Contraindication to CGM use, patient declines CGM use, or CGM not covered by patient's insurance;
* Concomitant use of other anti-diabetic medication (such as metformin); use of a short-acting insulin will not be considered an exclusion;
* Known or suspected fetal anomaly or aneuploidy;
* Prisoners;
* Ongoing prenatal care outside EVMS or planned delivery outside Sentara Norfolk General Hospital.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Weekly Time in Range | From Day 7 to Day 14 after study enrollment
  The mean blood glucose time in range as measured by the continuous glucose monitor

SECONDARY OUTCOMES:
Hypertensive disorders of pregnancy | From time of enrollment until time of delivery, up to 20 weeks following enrollment
  Development of hypertensive disorders of pregnancy
Preterm birth <34 weeks | From time of enrollment to 34 weeks gestation
  Delivery at less than 34 weeks gestation
Preterm birth <37 weeks | From time of enrollment until 37 weeks gestation
  Delivery prior to 37 weeks gestation
Spontaneous or Indicated Delivery | From time of enrollment until time of delivery, up to 20 weeks following enrollment
  Whether delivery was spontaneous or there was an indication for induction or cesarean delivery
Operative vaginal delivery | From time of enrollment to time of delivery, up to 20 weeks following enrollment
  Whether an operative vaginal delivery was indicated
Cesarean Delivery | From time of enrollment to time of delivery, up to 20 weeks following enrollment
  Whether a cesarean delivery was indicated
Estimated blood loss | Duration of labor, up to 24 hours
  The estimated blood loss during delivery
Quantitative blood loss | Duration of labor, up to 24 hours
  The quantified blood loss during delivery
Blood transfusion | From time of enrollment until hospital discharge (up to 42 days post-delivery)
  Whether a blood transfusion was necessary during or following delivery
Endometritis | From time of enrollment to hospital discharge (up to 42 days post-delivery)
  Incidence of endometritis (inflammation of uterine lining)
Chorioamnionitis | From time of enrollment until time of hospital discharge (up to 42 days post-delivery)
  Incidence of chorioamnionitis (placental and amniotic membrane infection)
Wound infection | From time of enrollment to hospital discharge (up to 42 days post-delivery)
  Infection of wounds left by labor
Venous thromboembolism | From time of enrollment to time of hospital discharge (up to 42 days post-delivery)
  Incidence of venous thromboembolism
Massive transfusion and postpartum hemorrhage | From time of enrollment until hospital discharge (up to 42 days post-delivery)
  Incidence of massive transfusion and postpartum hemorrhage
ICU admission | From time of enrollment until hospital discharge (up to 42 days post-delivery)
  Admission to the ICU
Maternal death | From time of enrollment to hospital discharge (up to 42 days post-delivery)
Antepartum death | From time of enrollment to time of delivery, up to 20 weeks following enrollment
  Fetal death
Intrapartum death | Duration of labor, up to 24 hours
  Fetal death during labor and delivery
Neonatal Intubation within 72 hours of birth | From time of delivery to 72 hours later
Continuous positive airway pressure (CPAP) within 72 hours of birth | From time of delivery to 72 hours later
  Use of CPAP for neonate within 72 hours of birth
High-flow nasal cannula (HFNC) within 72 hours of birth | From time of delivery to 72 hours later
Cardiopulmonary resuscitation within 72 hours of birth | From time of delivery to 72 hours later
Neonatal Hypoglycemia (glucose <35 mg/dL) requiring IV glucose therapy | From time of delivery to time of hospital discharge, up to 1 year following delivery
Birthweight | From time of delivery to time of hospital discharge, up to 1 year following delivery
  Infant birthweight
Neonatal encephalopathy | From time of delivery to time of hospital discharge, up to 1 year following delivery
Seizures | From time of delivery to time of hospital discharge, up to 1 year following delivery
  Incidence of neonatal seizures
Shoulder dystocia | From time of delivery to time of hospital discharge, up to 1 year following delivery
  Incidence of shoulder dystocia
Birth trauma | From time of delivery to time of hospital discharge, up to 1 year following delivery
  Incidence of neonatal birth trauma
Intracranial hemorrhage | From time of delivery to time of hospital discharge, up to 1 year following delivery
  Incidence of neonatal intracranial hemorrhage
Hyperbilirubinemia requiring phototherapy or exchange transfusion | From time of delivery to time of hospital discharge, up to 1 year following delivery
  Incidence of neonatal hyperbilirubinemia requiring phototherapy or exchange transfusion
NICU admission | From time of delivery to time of hospital discharge, up to 1 year following delivery
  Admission of neonate to the neonatal intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia 23507, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabbe SG, Calfas J, Simpson JL, et al. Obstetrics: Normal and Problem Pregnancies. Elsevier; 2017. doi:10.1016/C2013-0-00408-2
- [Background] Fishel Bartal M, Ashby Cornthwaite JA, Ghafir D, Ward C, Ortiz G, Louis A, Cornthwaite J, Chauhan SSP, Sibai BM. Time in Range and Pregnancy Outcomes in People with Diabetes Using Continuous Glucose Monitoring. Am J Perinatol. 2023 Apr;40(5):461-466. doi: 10.1055/a-1904-9279. Epub 2022 Jul 20. PMID 35858653
- [Background] Jethwani P, Saboo B, Jethwani L, Chawla R, Maheshwari A, Agarwal S, Jaggi S. Use of insulin glargine during pregnancy: A review. Diabetes Metab Syndr. 2021 Jan-Feb;15(1):379-384. doi: 10.1016/j.dsx.2021.01.012. Epub 2021 Jan 22. PMID 33540243
- [Background] Feghali M, Venkataramanan R, Caritis S. Pharmacokinetics of drugs in pregnancy. Semin Perinatol. 2015 Nov;39(7):512-9. doi: 10.1053/j.semperi.2015.08.003. PMID 26452316
- [Background] Eledrisi M, Suleiman NN, Salameh O, Khair Hamad M, Rabadi O, Mohamed A, Al Adawi R, Salam A. Twice-daily insulin glargine for patients with uncontrolled type 2 diabetes mellitus. J Clin Transl Endocrinol. 2018 Dec 11;15:35-36. doi: 10.1016/j.jcte.2018.12.002. eCollection 2019 Mar. No abstract available. PMID 30619716
- [Background] Ashwell SG, Gebbie J, Home PD. Twice-daily compared with once-daily insulin glargine in people with Type 1 diabetes using meal-time insulin aspart. Diabet Med. 2006 Aug;23(8):879-86. doi: 10.1111/j.1464-5491.2006.01913.x. PMID 16911626
- [Background] Lepore M, Pampanelli S, Fanelli C, Porcellati F, Bartocci L, Di Vincenzo A, Cordoni C, Costa E, Brunetti P, Bolli GB. Pharmacokinetics and pharmacodynamics of subcutaneous injection of long-acting human insulin analog glargine, NPH insulin, and ultralente human insulin and continuous subcutaneous infusion of insulin lispro. Diabetes. 2000 Dec;49(12):2142-8. doi: 10.2337/diabetes.49.12.2142. PMID 11118018
- [Background] Heinemann L, Linkeschova R, Rave K, Hompesch B, Sedlak M, Heise T. Time-action profile of the long-acting insulin analog insulin glargine (HOE901) in comparison with those of NPH insulin and placebo. Diabetes Care. 2000 May;23(5):644-9. doi: 10.2337/diacare.23.5.644. PMID 10834424
- [Background] Candido R, Wyne K, Romoli E. A Review of Basal-Bolus Therapy Using Insulin Glargine and Insulin Lispro in the Management of Diabetes Mellitus. Diabetes Ther. 2018 Jun;9(3):927-949. doi: 10.1007/s13300-018-0422-4. Epub 2018 Apr 13. PMID 29654514
- [Background] Westerbacka J, Duverne M, Grulovic N, Thummisetti S, Doder Z. Insulin glargine 300 U/mL safety data in pregnancy. Diabetes Obes Metab. 2025 May;27(5):2322-2325. doi: 10.1111/dom.16295. Epub 2025 Mar 19. No abstract available. PMID 40105254
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 201: Pregestational Diabetes Mellitus. Obstet Gynecol. 2018 Dec;132(6):e228-e248. doi: 10.1097/AOG.0000000000002960. PMID 30461693

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT07224893/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT07224893/ICF_001.pdf